CLINICAL TRIAL: NCT06881134
Title: Combinative Rehabilitation Strategy Combining Spatiotemporal Spinal Cord Stimulation and Real-time Triggering Exoskeleton (SCS-EXS) After Spinal Cord Injury: an Exploratory Study
Brief Title: Rehabilitation Combining Spatiotemporal Spinal Cord Stimulation and Real-time Triggering Exoskeleton After Spinal Cord Injury
Acronym: SCS-EXS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Wanru Duan, Associate Chief Physician, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024286001
Record Dates: First submitted 2024-12-03; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injury; Neuromodulation; Robot Assisted Gait Training
Keywords: motor recovery; limb dysfunction; neuromodulation; robot-assisted rehabilitation; machine interface
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SCS+EXS (Experimental): Eligible participants will undergo implantation of the spinal cord stimulation (SCS) system. Intraoperative electrophysiological monitoring will be used to adjust stimulation parameters. SCS will be tested postoperatively to assess the patient's tolerance to stimulation and its therapeutic effects. Parameters designed to improve sensory function and bladder/bowel control will be established. All parameters will be integrated into a sequential stimulation protocol. Additionally, the simultaneous activation of the SCS and the robotic exoskeleton will be tested to ensure smooth integration. Exoskeleton-assisted training will be conducted for no less than 1 hour per day (divided into two 30-minute sessions). Other rehabilitation interventions will be provided for at least 3 hours per day. Follow-ups will be conducted at 1, 2, 3, 6, and 12 months postoperatively.
  Interventions: Device: SCS+EXS

INTERVENTIONS:
Device: SCS+EXS — Eligible participants will undergo implantation of the spinal cord stimulation (SCS) system. Intraoperative electrophysiological monitoring will be used to adjust stimulation parameters. SCS will be tested postoperatively to assess the patient's tolerance to stimulation and its therapeutic effects. Parameters designed to improve sensory function and bladder/bowel control will be established. All parameters will be integrated into a sequential stimulation protocol. Additionally, the simultaneous activation of the SCS and the robotic exoskeleton will be tested to ensure smooth integration. Exoskeleton-assisted training will be conducted for no less than 1 hour per day (divided into two 30-minute sessions). Other rehabilitation interventions will be provided for at least 3 hours per day. Follow-ups will be conducted at 1, 2, 3, 6, and 12 months postoperatively.

SUMMARY:
Spinal cord injury (SCI) can be caused by trauma, inflammation, tumors, and other factors, often leading to issues such as impaired leg movement, abnormal sensation, and difficulties with bladder and bowel control. These challenges significantly affect the patient's quality of life. While there is currently no cure for spinal cord injury, the latest guidelines recommend spinal cord stimulation and robotic exoskeletons as effective rehabilitation methods.

Spinal cord stimulation (SCS) involves implanting a device that delivers electrical stimulations to aid in motor function recovery. Its safety and effectiveness have been proven in multiple clinical studies. For example, in 2022, a Swiss research team successfully helped three patients with severe spinal cord injuries regain the ability to stand, walk, and perform other movements, offering new hope for recovery.

A robotic exoskeleton is a wearable device that assists patients in movements like walking while promoting nerve and muscle recovery. This technology has become an increasingly important tool in spinal cord injury rehabilitation.

Recent studies have shown that combining spinal cord stimulation and robotic exoskeletons yields better outcomes. For instance, in 2023, an American research team demonstrated that after 24 weeks of combined therapy, patients could achieve independent walking or walk with the aid of assistive devices.

This study aims to combine spinal cord stimulation with robotic exoskeleton therapy to develop personalized rehabilitation plans for patients. The goal is to restore lower limb motor function and improve long-term quality of life.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) often results in long-term impairments in motor, sensory, and autonomic nervous functions, significantly reducing patients' quality of life and increasing the burden on families and society. Spinal cord stimulation (SCS) has emerged in recent years as a key therapeutic tool for functional rehabilitation following SCI. Multiple clinical research has confirmed its safety and effectiveness. Chalif et al. evaluated the applications of SCS in managing chronic SCI in a systematic review, highlighting its potential not only for motor function rehabilitation but also for improving bladder and bowel functions, regulating respiratory pressures, and enhancing gastrointestinal motility.

On the other hand, robotic exoskeleton as an innovative rehabilitation device, has demonstrated great potential in the treatment of SCI. By providing mechanical support, robotic exoskeletons assist patients in movement training, thereby promoting neural recovery and strengthening muscle function. Numerous clinical studies have investigated the benefits of exoskeleton training for lower limb rehabilitation in SCI patients, with results showing significant improvements in walking speed and independence. Future studies should explore the combination of exoskeleton training with other rehabilitation modalities to optimize outcomes and provide more robust clinical guidance.

The combination of SCS and robotic exoskeletons represents a novel direction in motor recovery for SCI. This approach aims to activate spinal neurons via SCS to restore muscle and neural functions, while robotic exoskeletons offer gait support and assist in motor activities, providing sensory feedback to construct a complete motor-sensory loop. This combination also holds promise for spinal circuit reorganization following SCI. Gorgey et al. reported three cases in 2020 and 2023 involving epidural spinal cord stimulation (eSCS) combined with exoskeleton training. The researchers identified optimal muscle activation parameters for walking and conducted 24 weeks of gait training with concurrent stimulation and exoskeleton use, achieving enhanced rehabilitation outcomes through this synergistic approach.

Currently, research on the combination of SCS and robotic exoskeletons for lower limb rehabilitation is limited. There is a lack of large-scale, long-term studies to validate the sustained efficacy of this combined approach. To address this gap, our study aims to develop an innovative rehabilitation system combining spatiotemporal spinal cord stimulation with real-time triggering exoskeleton. This research seeks to integrate the two systems clinically, assess their safety and effectiveness, and design personalized strategies to maximize patients' rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 14 and 65 years, with no restriction on gender;
* Diagnosed with spinal cord injury resulting in lower limb motor impairment due to trauma, inflammation, tumors, vascular diseases, iatrogenic factors, or other causes, confirmed through medical history, physical examination, and auxiliary tests;
* Diagnosed with spinal cord injury for at least 6 months, undergoing continuous routine rehabilitation for at least 1 month (including but not limited to physical therapy, acupuncture, hydrotherapy, etc., with daily training time ≥ 3 hours), but with no significant improvement in motor function over the past 2 months;
* Classified according to the ASIA impairment scale (AIS) based on the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), with an impairment grade of A, B, or C;
* Generally in good health, with an expected life expectancy of ≥ 12 months;
* The subject voluntarily agrees to participate in the study, signs an informed consent form, demonstrates good compliance, and is willing to cooperate with follow-up assessments.

Exclusion Criteria:

* Suffering from other diseases affecting lower limb muscle function besides spinal cord injury, including brain diseases (such as brain tumors, stroke, etc.), lower limb vascular diseases (such as lower limb vascular occlusion), peripheral nerve diseases, lower limb bone diseases (such as osteoarthritis, joint contractures, etc.);
* Congenital or acquired abnormalities in lower limb skeletal or muscular structure;
* Presence of surgical contraindications (such as adverse reactions to anesthesia, bleeding risks, or when the surgeon deems the patient unsuitable for surgery);
* Presence of active implanted devices, such as a pacemaker, defibrillator, drug infusion pump, cochlear implant, sacral nerve stimulator, etc. (whether turned on or off);
* Unable to undergo implantation of active devices due to treatment or examination requirements for other diseases;
* Suffering from severe cardiovascular diseases: ischemic heart disease or myocardial infarction of class II or higher, uncontrolled arrhythmias (including QTc interval ≥450 ms for males or ≥470 ms for females); heart failure of NYHA class III-IV, or echocardiogram showing left ventricular ejection fraction (LVEF) <50%;
* Coagulation dysfunction (INR >1.5 ULN or PT >ULN +4 seconds or APTT >1.5 ULN), bleeding tendency, or currently receiving thrombolytic or anticoagulant therapy;
* Severe infection within 4 weeks prior to surgery (such as requiring intravenous antibiotics, antifungals, or antivirals) or soft tissue infection in the lumbar or back region, or unexplained fever >38.5°C during screening or before surgery;
* Human Immunodeficiency Virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active pulmonary tuberculosis, active hepatitis B (HBV DNA ≥500 IU/ml), hepatitis C (positive hepatitis C antibody, and HCV-RNA levels above the detection threshold), or co-infection with both hepatitis B and C;
* Severe cerebrovascular events (including transient ischemic attacks, intracerebral hemorrhage, or ischemic stroke), deep vein thrombosis, or pulmonary embolism within 12 months prior to enrollment;
* Presence of metastatic malignant tumors or untreated malignant tumors;
* Major surgery or severe traumatic injury, fractures, or ulcers within 4 weeks prior to enrollment;
* Presence of addictive behaviors such as drug abuse or alcoholism;
* History of substance abuse of psychiatric drugs that cannot be discontinued, or presence of mental disorders;
* Pregnant women, breastfeeding women, women planning pregnancy, or women of childbearing age without reliable contraception;
* Presence of cognitive impairments or other factors preventing the patient from following treatment interventions and rehabilitation training;
* Situations that increase the risk associated with participation in the study or the study devices, and other conditions judged by the investigator that would make the patient unsuitable for inclusion in the study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall muscle strength improvement rate at 6 month | 6 month after combinative rehabilitation
  The overall muscle strength improvement rate is calculated as (Muscle strength at 6 month - Muscle strength at baseline) / Muscle strength at baseline.
  Muscle strength in the key muscles of both lower limbs will be assessed using the standard methods outlined in the ASIA Manual for Muscle Strength Testing. Scores will be assigned based on examination results on a scale from 0 to 5, while the anal sphincter will be scored as 0 or 1 depending on the presence or absence of contraction. The overall muscle strength is calculated as the total score of each muscle assessed.

SECONDARY OUTCOMES:
The overall muscle strength improvement rate at 1 month | 1 month after combinative rehabiliation
  The overall muscle strength improvement rate is calculated as (Muscle strength at 6 month - Muscle strength at baseline) / Muscle strength at baseline. Muscle strength in the key muscles of both lower limbs will be assessed using the standard methods outlined in the ASIA Manual for Muscle Strength Testing. Scores will be assigned based on examination results on a scale from 0 to 5, while the anal sphincter will be scored as 0 or 1 depending on the presence or absence of contraction. The overall muscle strength is calculated as the total score of each muscle assessed.
The overall muscle strength improvement rate at 2 month | 2 month after combinative rehabilitation
  The overall muscle strength improvement rate is calculated as (Muscle strength at 6 month - Muscle strength at baseline) / Muscle strength at baseline. Muscle strength in the key muscles of both lower limbs will be assessed using the standard methods outlined in the ASIA Manual for Muscle Strength Testing. Scores will be assigned based on examination results on a scale from 0 to 5, while the anal sphincter will be scored as 0 or 1 depending on the presence or absence of contraction. The overall muscle strength is calculated as the total score of each muscle assessed.
The overall muscle strength improvement rate at 3 month | 3 month after combinative rehabilitation
  The overall muscle strength improvement rate is calculated as (Muscle strength at 6 month - Muscle strength at baseline) / Muscle strength at baseline. Muscle strength in the key muscles of both lower limbs will be assessed using the standard methods outlined in the ASIA Manual for Muscle Strength Testing. Scores will be assigned based on examination results on a scale from 0 to 5, while the anal sphincter will be scored as 0 or 1 depending on the presence or absence of contraction. The overall muscle strength is calculated as the total score of each muscle assessed.
The overall muscle strength improvement rate at 12 month | 12 month after combinative rehabilitation
  The overall muscle strength improvement rate is calculated as (Muscle strength at 6 month - Muscle strength at baseline) / Muscle strength at baseline. Muscle strength in the key muscles of both lower limbs will be assessed using the standard methods outlined in the ASIA Manual for Muscle Strength Testing. Scores will be assigned based on examination results on a scale from 0 to 5, while the anal sphincter will be scored as 0 or 1 depending on the presence or absence of contraction. The overall muscle strength is calculated as the total score of each muscle assessed.
Assisted standing time | 6 month after combinative rehabiliation
  The maximum standing time that the subject can maintain with minimal orthotic or manual assistance (in minutes).
6-minute walking test | 6 month after combinative rehabiliation
  In a 30-meter straight corridor, mark every 3 meters. Instruct the subject to walk back and forth along the corridor as quickly as possible without hesitation or pausing when turning. Measure the maximum walking distance (in meters) covered within 6 minutes. If the subject experiences shortness of breath or fatigue, they may slow down or rest, resuming walking as soon as symptoms improve. If chest tightness, chest pain, or any other discomfort occurs, the subject should inform the tester immediately. If the subject is unable to walk, record the result as NA.
10-meter walking test | 6 month after combinative rehabiliation
  In a straight corridor at least 14 meters long, mark the 0, 2, 12, and 14-meter points. Instruct the subject to walk from the 0-meter mark to the 14-meter mark. Record the time taken for the toes to pass from the 2-meter mark to the 12-meter mark. Calculate the walking speed (in meters per second) by dividing 10 meters by the recorded time.
  The subject may choose to walk at a comfortable pace or at maximum effort, but the selected pace should be clearly documented in the record. If the subject is unable to walk, record the result as NA.
Spinal Cord Injury Walking Index | 6 month after combinative rehabiliation
  The subject is rated according to the standards provided by the Spinal Cord Injury Walking Index.
Gait parameters | 6 month after combinative rehabiliation
  The parameters are evaluated based on the gait analysis provided by the robotic exoskeleton, for example, stride length, step height, cycle, walking speed, etc.
Pain level | 6 month after combinative rehabiliation
  According to the Visual Analog Scale (VAS), which consists of a 100mm line, one end represents "no pain at all," and the other end represents "the most intense pain imaginable" or "pain at its extreme." The subject is asked to mark the position on the line that corresponds to the intensity of pain they are currently experiencing.
Quality of Life Scale | 6 month after combinative rehabiliation
  The Health Survey Questionnaire consists of 9 dimensions and 36 items, measuring 8 aspects of health: physical functioning (PF), role limitations due to physical health (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH).
Electromyography parameters | 6 month after combinative rehabiliation
  Nerve conduction velocity of the peroneal nerve and tibial nerve.
Urodynamic parameters | 6 month after combinative rehabiliation
  Post-void residual volume, maximum free flow rate, and bladder compliance volume.
Functional MRI | 6 month after combinative rehabiliation
  Spinal cord functional MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China